CLINICAL TRIAL: NCT02718001
Title: Edwards EVOQUE Eos Mitral Valve Replacement: Investigation of Safety and Performance After Mitral Valve Replacement With Transcatheter Device (MISCEND)
Brief Title: Edwards EVOQUE Eos MISCEND Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-05C
Record Dates: First submitted 2016-03-01; First posted 2016-03-24 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
Keywords: Mitral; Regurgitation; Insufficiency; Degenerative; Functional; Primary; Secondary; Organic; Transcatheter; TMVR; TMVI; Heart Valve; Mitral Valve; Transseptal; Trans-Septal; Transeptal; Severe
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux; Neoplasm Metastasis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the Edwards EVOQUE Eos mitral valve replacement system
  Interventions: Device: Edwards EVOQUE Eos Mitral Valve Replacement System

INTERVENTIONS:
Device: Edwards EVOQUE Eos Mitral Valve Replacement System — Replacement of the mitral valve through a transcatheter approach
  Other Names: CardiAQ-Edwards™ Transcatheter Mitral Valve (TMV); Edwards FORTIS™ Transcatheter Mitral Valve (TMV); Transcatheter Mitral Valve Replacement (TMVR); Edwards EVOQUE Transcatheter Mitral Valve Replacement System

SUMMARY:
Study to evaluate the safety and performance of the Edwards EVOQUE Eos mitral valve replacement system

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-arm, and non-randomized study designed to evaluate the safety and performance of the Edwards EVOQUE Eos mitral valve replacement system.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant, symptomatic mitral regurgitation
* High risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Patient is inoperable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2015-02-06 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse events | 30 days
  Proportion of patients with major adverse events

SECONDARY OUTCOMES:
NYHA functional class | 30 days, 6 Months, 12 Months, annual for five years
  Number of patients with improvement in NYHA class
Six minute walk test | 30 days, 6 Months, 12 Months, annual for five years
  Increase in distance (m) from baseline
Reduction in MR grade | 30 days, 6 Months, 12 Months, annual for five years
  Number of patients with reduction in MR grade from baseline
Device Success | Immediately after procedure
  Proportion of patients with device deployed as intended and delivery system successfully retrieved
Procedural Success | Discharge or 7 days post-procedure, whichever occurs first
  Proportion of patients with device success without significant paravalvular leak
Clinical Success | 30 days
  Proportion of patients with procedural success without major adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA
Locations (19):
- United States (16):
  - Sutter Mills-Peninsula, Burlingame, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Emory University Hospital/Emory University Hospital Midtown, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Morristown Medical Center, Morristown, New Jersey
  - St. Francis Hospital, Roslyn, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston/Memorial Hermann Texas Medical Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec-Université Laval, Québec
  - St. Michael's Hospital, Toronto

IPD SHARING:
Plan to Share IPD: No